CLINICAL TRIAL: NCT06804564
Title: Comparative Effectiveness of Cold and Warm Water Immersion in Mitigating Delayed Onset Muscle Soreness: a Multi-Arm Randomized Controlled Trial
Brief Title: Cold Vs Warm Water Immersion for DOMS Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKE 01-80/2023
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Sham Comparator): Participants subjected only to standard biomechanical, functional, and blood measurements, without the use of regenerative therapies.
  Interventions: Other: Simulated Laser Therapy
- Cold Water Immersion (CWI) (Experimental): Participants are subjected to a bath in cold water (10-12°C) for 10 minutes with the lower limbs submerged to waist height.
  Interventions: Other: Cold Water Immersion (CWI)
- Hot Water Therapy (HOT) (Experimental): Immersing the whole body in hot (40°C) water.
  Interventions: Other: Hot Water Immersion (HWI)

INTERVENTIONS:
Other: Cold Water Immersion (CWI) — Standard immersion baths with temperature monitoring and ice supplementation. Lower limbs immersed up to the hip. Water temperature maintained at 10-12°C. Duration: 15 minutes per session. Participants perform active ankle flexion/extension to promote circulation.
  Other Names: cryotherapy
  Arms: Cold Water Immersion (CWI)
Other: Hot Water Immersion (HWI) — Controlled immersion baths. Lower limbs immersed up to the hip. Water temperature maintained at 40°C. Duration: 15 minutes per session.
  Arms: Hot Water Therapy (HOT)
Other: Simulated Laser Therapy — Deactivated low-level laser therapy (LLLT) device. Applicator positioned over quadriceps muscle belly. Duration: 15 minutes, with no active laser output to simulate treatment conditions.
  Arms: Control group

SUMMARY:
The study investigates the effectiveness of physical strategies in addressing Delayed Onset Muscle Soreness (DOMS) in physically active individuals. DOMS, a common phenomenon following intense or novel physical activity, is characterized by pain, inflammation, and functional impairments such as reduced range of motion, muscle strength, and endurance. These symptoms peak between 24-72 hours post-exercise and are attributed to micro-damage in muscle and connective tissue, followed by inflammatory responses. Despite extensive research, the efficacy of various therapeutic interventions remains inconclusive due to heterogeneity in study designs, outcome measures, and quality of evidence.

The primary objective of this study is to systematically assess and compare the effectiveness of cold water immersion (CWI) or hot water immersion (HWI), in mitigating DOMS symptoms. This study will utilize a multi-arm, parallel, randomized controlled trial (RCT) design to evaluate therapeutic outcomes against a control group receiving simulated therapy.

By employing a standardized exercise protocol to induce DOMS and unified assessment methodologies (e.g., biomechanical, biochemical, and functional tests), the study aims to provide robust evidence for the efficacy of these interventions. The findings will contribute to optimizing post-exercise recovery strategies, offering reliable therapeutic protocols for both clinical and athletic settings.

DETAILED DESCRIPTION:
The study is a multi-arm, parallel, randomized controlled trial (RCT) designed to evaluate the effectiveness of cold water immersion (CWI), warm water immersion (WWI), and simulated laser therapy (control group) in mitigating Delayed Onset Muscle Soreness (DOMS). This trial aims to compare the physiological, biochemical, and functional outcomes of these interventions following exercise-induced muscle damage in healthy male participants. DOMS, which arises from eccentric physical activities, presents with symptoms such as muscle pain, stiffness, inflammation, and functional limitations, reaching a peak 24-72 hours post-exercise.

Setting and Duration The study will be conducted at the laboratories of the Faculty of Physical Education and Health at AWF Biała Podlaska between March and May 2024. The laboratory sessions will take place on weekdays from 8:00 AM to 4:00 PM.

Methodology Participants will be randomly assigned to one of three study groups

Cold Water Immersion (CWI):

Participants will submerge their lower limbs in water maintained at 10-12°C for 15 minutes. The water temperature will be regulated with ice additions to ensure consistency. Participants will perform light movements, such as ankle flexion and extension, to stimulate blood flow.

Sessions will occur 1 hour post-exercise, and at 24 and 48 hours.

Hot Water Immersion (HWI):

Participants will immerse their lower limbs in water at 40°C for 15 minutes, maintaining consistent temperature conditions.

Sessions will follow the same schedule as the CWI group (1, 24, and 48 hours post-exercise).

Simulated Laser Therapy (Control Group):

Participants in this group will receive simulated low-level laser therapy (LLLT). A deactivated laser device will be positioned over the muscles to mimic therapy without delivering actual treatment. Simulated sessions will align with the intervention schedule of the other groups.

Study Procedure

The study comprises three phases:

Baseline Measurements (Phase 1):

Conducted in the morning, fasting, followed by standardized functional and biomechanical tests two hours after a light meal.

Measurements include body composition, joint range of motion, muscle stiffness (elastography), pain assessments (VAS scale), and venous blood sampling to measure baseline biochemical markers.

Exercise-Induced Muscle Damage (Phase 2):

Participants will perform eccentric exercises designed to induce DOMS, targeting the quadriceps muscles. The exercise protocol includes five sets of 20 drop jumps from a 60 cm height with a 5-minute rest between sets.

Experienced physiotherapists will ensure the correct execution of exercise.

Post-Exercise Monitoring and Intervention (Phase 3):

Interventions (CWI, WWI, or simulated LLLT) will be administered within an hour post-exercise and repeated at 24 and 48 hours.

Functional tests and blood sampling will be conducted pre-intervention and at 24, 48, 72, and 96 hours post-exercise to assess recovery dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-25 years
* BMI between 18.5 and 30 kg/m²
* Experiencing muscle pain (VAS scale) > 5 for muscle soreness within 12 to 30 hours post-exercise
* Engage in moderate physical activity 2-5 hours/week, according to the International Physical Activity Questionnaire-Short Form (IPAQ-SF).
* They must voluntarily sign a written informed consent approved by an ethics/bioethics committee after sufficient explanation prior to participating in the study.

Exclusion Criteria:

* Inflammatory diseases within the past 6 months
* Neurological disorders that affect muscle strength
* Ongoing use of steroids, analgesics, muscle relaxants, or other medications deemed inappropriate by the researchers, including antispasmodics, antidepressants, antidiarrheals, antibiotics, or thrombolytics
* Unstable medical condition such as cardiovascular disease, respiratory disease, gastrointestinal disease, hepatobiliary disease, metabolic disease, endocrine disease, kidney disease, urinary tract disease, genetic disorders, or issues related to the nervous system or mental health.
* Participants who have abused alcohol or drugs in the past year, do not wish to follow the study guidelines, or are deemed inappropriate for the study by the researcher will also be excluded.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Soreness (VAS Score) | Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours)
  Muscle Soreness Measured by the Visual Analog Scale (0-10) Description: The Visual Analog Scale (VAS) ranges from 0 ("no muscle pain") to 10 ("worst possible pain"). Higher scores indicate a worse outcome (greater pain).

SECONDARY OUTCOMES:
Change in Biochemical Markers of Muscle Damage (Creatine Kinase) | Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours)
  Blood samples will be collected at baseline, 24 h, 48 h, and 72 h post-exercise and analyzed for serum Creatine Kinase (U/L) using standard immunoassay methods.
Change in Quadriceps Muscle Strength (Nm) measured by Dynamometer at Baseline, 24h, 48h, 72h Post-Exercise | Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours)
Change in Quadriceps Muscle Tissue Elasticity (kPa) measured by Ultrasound Elastography at Baseline, 24h, 48h, 72h Post-Exercise | Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours)
Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours) | Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours)
Change in Biochemical Markers of Muscle Damage: Myoglobin | Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours)
  Blood samples will be collected at baseline, 24 h, 48 h, and 72 h post-exercise and analyzed for Myoglobin (ng/mL), using standard immunoassay methods.
Change in Inflammation markers (IL-6, TNF-α) | Baseline to 72 hours post-exercise, with measurements at Day 1 (24 hours), Day 2 (48 hours), and Day 3 (72 hours)
  Blood samples will be collected at baseline, 24 h, 48 h, and 72 h post-exercise and analyzed for Interleukin 6 (IL-6) and Tumor Necrosis Factor α (TNF-α) (pg/mL), using standard immunoassay methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Akademia Wychowania Fizycznego w Warszawie, Biała Podlaska, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Because the study sample is small and participants were locally recruited, there is a heightened risk that individual identities could be inferred. Therefore, we do not plan to share de-identified participant data in order to protect privacy and confidentiality.